CLINICAL TRIAL: NCT07318714
Title: A Phase 1/2 Multicenter, Open-label, Dose Escalation Study Followed by a Randomized, Double-blind Sham-controlled Dose Expansion Study to Evaluate the Safety, Tolerability and Efficacy of ASP2246 in Adult Participants Who Have Motor Dysfunction Associated With Late Subacute to Chronic Ischemic Stroke Due to Supratentorial Perforator Area Infarction
Brief Title: A Study of ASP2246 for People Who Have Movement Problems Caused by Brain Injury After a Stroke
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2246-CL-0101
Record Dates: First submitted 2026-01-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Ischemic Stroke
Keywords: Safety; Tolerability; Efficacy; ASP2246
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ASP2246 Dose Escalation (Part 1) (Experimental): Participants will undergo stereotactic brain surgery and receive sequential dose levels of a single intracerebral parenchymal infusion of ASP2246. Participants will undergo rehabilitation therapy.
  Interventions: Drug: ASP2246; Procedure: Brain surgery; Other: Rehabilitation therapy
- ASP2246 Dose Expansion (Part 2) (Experimental): Participants will undergo stereotactic brain surgery and receive a single intracerebral parenchymal infusion of ASP2246. The dosage will be selected from Dose Escalation (Part 1). Participants will undergo rehabilitation therapy.
  Interventions: Drug: ASP2246; Procedure: Brain surgery; Other: Rehabilitation therapy
- Sham Dose Expansion (Part 2) (Sham Comparator): Participants will undergo a sham surgery and rehabilitation therapy.
  Interventions: Procedure: Sham surgery; Other: Rehabilitation therapy

INTERVENTIONS:
Drug: ASP2246 — Intracerebral parenchymal infusion via SmartFlow Neuro cannula.
  Arms: ASP2246 Dose Escalation (Part 1); ASP2246 Dose Expansion (Part 2)
Procedure: Brain surgery — Stereotactic brain surgery
  Arms: ASP2246 Dose Escalation (Part 1); ASP2246 Dose Expansion (Part 2)
Procedure: Sham surgery — Sham surgery without the dura incised.
  Arms: Sham Dose Expansion (Part 2)
Other: Rehabilitation therapy — Rehabilitation 3 days per week for up to 12 weeks.

SUMMARY:
This study is for adults who have difficulty moving a few months after a stroke. In this study, ASP2246 will be given to people for the first time. This is known as a "first in human" study.

The main aims of the study are to check the safety of ASP2246, how well people tolerate it, and to find suitable doses of ASP2246 to use later in this study and in future studies.

This study has 2 parts. In Part 1, people will have brain surgery. During the surgery, different small groups of people will receive a lower to a higher dose of ASP2246. Each dose will be given slowly through a special tube to the damaged part of the brain (intracerebral parenchymal infusion). Any medical problems will be recorded at each dose. This is done to find suitable doses to use in Part 2 of the study.

In Part 2, other different groups of people will undergo the same type of brain surgery. Some people will receive a higher dose of ASP2246, and some people will receive a lower dose of ASP2246. These are the doses from Part 1. Also, another group of people won't be given ASP2246 during brain surgery. This is known as a sham procedure. This is done so neither the people taking part in Part 2, nor the study doctors (apart from the surgeons) know who will be given ASP2246.

After brain surgery, people will be observed for about 2 weeks. After this, they will have physical therapy and continue to have safety checks for about 1 year after their brain surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant should have had an ischemic cerebral infarction at least 3 months, but not more than 12 months, before signing informed consent. This stroke must be the first-ever stroke for the participant.
* Participant has current neuromotor dysfunction with a modified Rankin Scale (mRS) score between 2 to 4 at screening.
* Participant has Fugl-Meyer Assessment (FMA)- upper extremity (UE) score ≥ 20 to ≤ 50 and FMA-lower extremity (LE) score < 21 at screening.
* Participant has supratentorial perforator area infarction (single lacunar infarction or branch-atheromatous disease [BAD]), as assessed clinically and by magnetic resonance imaging (MRI) at screening.
* Participant has completed recovery phase rehabilitation after cerebral infarction and spontaneous improvement is not expected during the study period.
* Participant is willing and physically able to participate in the designated rehabilitation therapy during the study period.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woma(e)n of childbearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test at screening (Unique to Japan: with a medical interview) and agrees to follow contraceptive guidance from the time of giving informed consent to at least 180 days after surgery.
* Female participant must not be breastfeeding or lactating starting at screening and for 180 days after surgery.
* Female participant must not donate ova after undergoing surgery and for 180 days after surgery.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) for a minimum of 180 days after surgery.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for a minimum of 180 days after surgery.
* Male participant must not donate sperm for a minimum of 180 days after surgery.
* Participant agrees not to participate in another interventional study (including rehabilitation) while receiving study intervention/participating for up to 52 weeks in the present study.
* Participant agrees that the use of antiplatelet, oral anticoagulant or nonsteroidal anti-inflammatory drugs (NSAIDs) will be determined by the local medical staff in accordance with the American College of Chest Physicians Clinical Pharmacy 2022 Guidelines and the Japanese Guidelines for the Management of Stroke 2021. The Japanese guidelines specify that no antiplatelet, oral anticoagulant or NSAIDs are to be restarted post-surgery until results of the day 1 head MRI or computerized tomography (CT) are reviewed and restarting medication is deemed safe.

Exclusion Criteria:

* Participant has a cerebral infarct volume > 3.4 cm^3 or < 0.37 cm^3, as measured by MRI (use of either a central or local reading is acceptable).
* Participant has a primary intracerebral or intracranial hemorrhage.
* Participant has a history of central nervous system (CNS) malignancy or a known presence of any malignancy, unless in remission for > 5 years. Exception: The participant with basal or squamous cell skin cancer that has been successfully treated will be considered eligible even if they have been in remission for < 5 years.
* Participant had motor dysfunction of mRS > 2 before the onset of the stroke (premorbid mRS).
* Participant has a history of seizures.
* Participant has apparent contractures impeding joint movement at shoulder, elbow, forearm, wrist, hand, hip, knee or ankle.
* Participant with spasticity of grade 2 or higher on the modified Ashworth Scale.
* Participant has any other neurologic, neuromuscular or orthopedic disease that limits motor function.
* Participant has an active infection.
* Participant has a history of or current diagnosis of immunodeficiency.
* Participant has been deemed to have a high risk of recurrent stroke during the study period (e.g., a family history strongly suggestive of hereditary cerebrovascular disease, such as moyamoya disease and cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy).
* Participant has an uncontrolled systemic illness, including, but not limited to, hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 95 mmHg), resistant hypertension (systolic blood pressure [BP] ≥ 140 mmHg or diastolic BP ≥ 90 mmHg in a participant who is taking 3 or more medications for hypertension), bleeding disorders, hypercoagulability, diabetes, renal, hepatic or cardiac failure, morbid obesity, or uncontrolled sleep apnea.
* Participant has any positive findings on tests for occult malignancy, unless a nonmalignant etiology is confirmed.
* Participant has an uncontrolled major psychiatric illness, including depression (Hamilton Score of > 14).
* Participant has a presence of craniectomy (without bone flap replacement) or other contraindication for stereotactic surgery.
* Participant has signs and symptoms of intracranial herniation or increased intracranial pressure.
* Participant with a history of, or electrocardiogram (ECG) evidence suggestive of, recent myocardial infarction (within 6 months of surgery), major dysrhythmia, atrial fibrillation or congestive heart failure.
* Participant has a substance-related and addictive disorders as defined by the Diagnostic and Statistical Manual of Mental Disorders-5 criteria, including drug or alcohol use.
* Participant has contraindications to MRI or MRI contrast agent(s).
* Participant has Montreal Cognitive Assessment (MoCA) score < 26.
* Participant has a history of suicide attempt(s), suicidal behavior, or suicidal ideation (indicated by a 'yes' response to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale [C-SSRS]) within 12 months prior to study enrollment, or who is assessed at screening to be at a significant risk of committing suicide.
* Participant has a history of using warfarin or direct oral anticoagulant (DOAC). Exception: The participant will be considered eligible if the medication was discontinued at least 6 months prior to study enrollment, and the embolic source has resolved without recurrence.
* Participant has a history of neuroleptic drug use. Exception: The participant will be considered eligible if they are neuroleptic medication-free for at least 6 months and their psychiatric symptoms remain mild, stable and do not meet the exclusion criteria.
* Participant has a history of antiepileptic drug use for seizures. Note: For the participant who has used or is using antiepileptic medications for conditions other than seizures, a detailed risk assessment needs to be conducted to determine eligibility.
* Participant has had botulinum toxin injection, phenol injection, intrathecal baclofen, or any other interventional treatments for spasticity (except bracing and splinting) within the previous 3 months.
* Participant has present or previous history of participation in a study with ASP2246.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has inadequate organ function as indicated by the laboratory values at screening.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has known or suspected hypersensitivity to ASP2246 or any components of the formulation used.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-Limiting Toxicity (DLT) | Up to 2 Weeks
  A DLT will be defined as an Adverse Event (AE) ≥ 3 Grade that is attributed to study intervention or surgical procedure. This determination will be based on the investigator's initial assessment of causality and will be confirmed by the Dose Escalation and Safety Committee (DESC). A Grade 3 AE is defined as a severe or medically significant event that is not immediately life-threatening, but may cause hospitalization or prolongation of hospitalization, be disabling, or limit a patient's ability to perform self-care activities of daily living (ADL).
Number of participants with Treatment-Emergent Adverse Events (TEAEs) | Up to 52 Weeks
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
  A TEAE is defined as an AE observed until 52 weeks after surgery on day 1.
Number of participants with Serious Adverse Events (SAEs) | Up to 52 Weeks
  A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or other situations.
Number of participants with an Adverse Event of Special Interest (AESI) | Up to 52 Weeks
  An AESI includes intracranial hemorrhage, cerebral edema (local or extensive), meningitis/encephalitis/encephalopathy (infectious or aseptic), seizures, worsening or new onset of neurologic deficits, intracranial malignancies/tumor formation, and immunogenic reactions.
Number of Participants with Suicidal Ideation and/or Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 52 Weeks
  The C-SSRS is a validated, clinician-administered tool used to assess suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) will be reported.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP2246 in whole blood: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 52 Weeks
  AUCinf will be recorded from the PK whole blood samples collected.
PK of ASP2246 in whole blood: AUC from the time of dosing up to the time of the last measurable concentration (AUClast) | Up to 52 Weeks
  AUClast will be recorded from the PK whole blood samples collected.
PK of ASP2246 in whole blood: maximum concentration (Cmax) | Up to 52 Weeks
  Cmax will be recorded from the PK whole blood samples collected.
PK of ASP2246 in plasma: AUCinf | Up to 52 Weeks
  AUCinf will be recorded from the PK plasma samples collected.
PK of ASP2246 in plasma: AUClast | Up to 52 Weeks
  AUClast will be recorded from the PK plasma samples collected.
PK of ASP2246 in plasma: Cmax | Up to 52 Weeks
  Cmax will be recorded from the PK plasma samples collected.
Number of participants with anti-polyethylene glycol (PEG) antibodies | Up to 52 Weeks
  Anti-PEG antibody status will be recorded from the serum samples collected.
Number of participants with anti-neurogenic differentiation 1 transcription factor (NeuroD1) antibodies | Up to 52 Weeks
  Anti-NeuroD1 antibody status will be recorded from the serum samples collected.
Change from baseline in proinflammatory cytokine response | Baseline and up to Day 8
  Proinflammatory cytokine response will be recorded from the serum samples collected.
Change from baseline in complement activation | Baseline and up to Day 8
  Complement activation will be recorded from the serum samples collected.
Change from baseline in Fugl-Meyer Assessment (FMA) (motor function) total score | Baseline, Week 24 and Week 52
  The FMA consists of five domains: motor function, sensory function, balance, joint range of motion, and joint pain, evaluating a total of 155 items. In this study, only the motor function score will be utilized to capture motor-specific changes. The motor function score ranges from 0 (hemiplegia) to 100 points (normal motor function), combing scores from upper extremity (UE) assessment and lower extremity (LE) assessment.
Change from baseline in FMA-UE total score | Baseline, Week 24 and Week 52
  FMA-UE evaluates movements of the shoulder, elbow, forearm, wrist, hand as well as coordination and reflex actions.
Change from baseline in FMA-LE total score | Baseline, Week 24 and Week 52
  FMA-LE evaluates movements of the hip, knee, ankle as well as coordination and reflex actions.
Number of participants with decrease of at least 1 point from baseline in modified Rankin Scale (mRS) score | Baseline, Week 24 and Week 52
  The mRS ranges from 0 (no symptoms) to 6 (deceased), capturing levels of disability from full independence to severe dependence.
Change from baseline in mRS score | Baseline, Week 24 and Week 52
  The mRS ranges from 0 (no symptoms) to 6 (deceased), capturing levels of disability from full independence to severe dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Inc

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/